CLINICAL TRIAL: NCT01574625
Title: Post-Approval Study for the MOSAIC® Bioprostheses: A Long Term Follow Up Study.
Brief Title: Post-Approval Study for the MOSAIC® Bioprostheses
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: MOSAIC
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Stenosis and/or Insufficiency; Mitral Valve Stenosis and/or Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mosaic prosthetic heart valve: All patients who were enrolled and implanted with a Mosaic bioprosthesis in the Albertinen-Krankenhaus (Hamburg, Germany) during the previous Mosaic PMA study and who agree to participate in this long-term follow-up study by informed consent.

SUMMARY:
A Single Center Non-Interventional Post-Market Release, Long Term Follow Up study of patients who underwent Isolated Aortic Valve Replacement or Isolated Mitral Valve Replacement with a Medtronic Mosaic Bioprosthesis. The purpose of this study is to evaluate the long term safety, efficacy and clinical performance of the Mosaic Bioprostheses.

DETAILED DESCRIPTION:
Objectives:

The primary objectives of this study are to evaluate the long-term safety, efficacy and clinical performance.

Study Design:

This is a prospective, single center, non-interventional, non-randomized, post-market release clinical study

Sample Size and Study Duration:

A total of 255 patients had aortic valve replacement and 47 patients had mitral valve replacement in the Albertinen-Krankenhaus (Hamburg, Germany) during the previous Mosaic Pre-Market approval (PMA) study.

All surviving patients from the Mosaic Pre-Market Approval study at this center, will be invited to participate. Approximately 225 patients will be invited.

This study is intended to serve as an ongoing source of information on long-term durability and safety of the CE-marked Medtronic Mosaic bioprosthesis. As such the study is to continue indefinitely until the last follow-up visit (until patient study exit due to patient death, withdrawal of patient consent,...) of the last study patient.

PATIENT SELECTION:

Inclusion criteria:

* All patients who were enrolled and implanted with the Mosaic bioprosthesis in the Albertinen-Krankenhaus (Hamburg, Germany) during the previous Mosaic PMA study, will be invited to participate in this long- term follow-up study.
* Patients who are able to provide informed consent

Exclusion criteria:

* Patients who are not from the Albertinen-Krankenhaus (Hamburg, Germany) and who did not participate in the Mosaic PMA study are ineligible for this study.
* Patients refusing or not able to provide informed consent.
* Patients not willing and unable to comply with the Clinical Investigation Plan (CIP)-requirements.

Data Requirements and analysis:

For each patient enrolled in the study, information will be collected annually. Data will be collected on the patient status and device hemodynamic performance by echocardiography. Patient identity is anonymized.

Appropriate statistical analysis will be performed for the collected clinical data.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were enrolled and implanted with a Mosaic bioprosthesis in the Albertinen-Krankenhaus (Hamburg, Germany) during the previous Mosaic PMA study, will be invited to participate in this long-term follow- up study.
* Patients who are able to provide informed consent

Exclusion Criteria:

* Patients who are not from the Albertinen-Krankenhaus (Hamburg, Germany) and who did not participate in the Mosaic PMA study are ineligible for this study.
* Patients refusing or not able to provide informed consent.
* Patients not willing and unable to comply with the CIP-requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population for this study includes all patients who were enrolled and implanted with a Mosaic bioprosthesis in the Albertinen-Krankenhaus (Hamburg, Germany) during the previous Mosaic PMA study and who are still available for follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2001-04; Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
long-term safety of the valve | Long term follow up: 10 years and longer
  The long-term safety of the valve will be assessed by the rate of valve related complications.
The long-term durability of the valve will be assessed by measuring hemodynamic performance of the valve Long-term performance of the valve | Long term follow up: 10 years and longer
  The long-term performance of the valve will be assessed by measuring hemodynamic performance of the valve by echo
Long-term efficacy of the valve | Long term follow up: 10 years and longer
  The long-term efficacy of the valve will be assessed by evaluating the New York Heart Association Functional Classification (NYHA)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Christian Rieß, Prof. Dr., Principal Investigator — Albertinen Krankenhaus
Locations (1):
- Albertinen Krankenhaus, Hamburg, Germany

REFERENCES:
- [Result] Riess FC, Cramer E, Hansen L, Schiffelers S, Wahl G, Wallrath J, Winkel S, Kremer P. Clinical results of the Medtronic Mosaic porcine bioprosthesis up to 13 years. Eur J Cardiothorac Surg. 2010 Jan;37(1):145-53. doi: 10.1016/j.ejcts.2009.04.073. Epub 2009 Aug 19. PMID 19695889
- See also: General Medtronic website — http://www.medtronic.com